CLINICAL TRIAL: NCT01911481
Title: Maternal Oral Hydration and External Cephalic Version: a Single Blind Randomised Controlled Trial
Brief Title: Maternal Oral Hydration and External Cephalic Version
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: IDRI
Record Dates: First submitted 2013-07-22; First posted 2013-07-30 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: External Cephalic Version; Maternal Oral Hydration

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hydration (Experimental): after recruitment the women in hydration group will be invited to drink 2 litres of water,in 2 hours
  Interventions: Other: hydration
- control (No Intervention)

INTERVENTIONS:
Other: hydration
  Arms: hydration

SUMMARY:
The investigators are carrying out a study of 164 pregnant women, with breech presentation at term who will undergo to external cephalic version. The investigators' goal is to know if oral maternal hydration can increase the successful of external cephalic version

ELIGIBILITY:
Inclusion Criteria:

* single gestation
* breech presentation
* from 37 to 41,5 weeks
* without pregnancy complications
* fetus adequate for gestational age
* without fetal malformations
* intact membranes
* amniotic fluid index between 7 and 24 cm
* placenta properly inserted

Exclusion Criteria:

* age less than 18 years
* maternal disease at risk of fluid overload (cardiac disease, renal impairment, moderate or severe preeclampsia or hypertension and diabetes)
* contraindications for vaginal birth
* vaginal blood loss
* uterine contractions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2011-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with external cephalic version successful after maternal oral hydration | The primary outcome will be assessed by ultrasound examination, 5 minutes after ending of the external cephalic version
  The primary outcome of the study is to evaluate the successful rate of external cephalic version, after oral intake of two litres of water

SECONDARY OUTCOMES:
amniotic fluid volume | 1 hour after the end of oral maternal hydration (2 litres)
  We will assess the amniotic fluid index at recruitment (Baseline). 1 hour after ending of oral intake (2 litres of water), we will revalue the amniotic fluid volume
type of birth | at birth
  We will record if the woman will give birth by cesarean section or vaginal birth (spontaneous or operative)

OTHER OUTCOMES:
type of breech presentation | Baseline
  At recruitment we will assess the type of breech (frank breech, complete breech, footling or incomplete breech)
placental localisation | baseline
  At recruitment we will assess the placental localisation (anterior, posterior, right lateral, left lateral or fundal)
foetal back position | baseline
  At recruitment we will evaluate the position of fetal back (anterior, posterior, right or left lateral)

CONTACTS AND LOCATIONS:
Overall Officials: Antonietta A Scian, MD, Study Chair — San Gerardo Hospital
Locations (1):
- San Gerardo Hospital, Monza, Monza Brianza, Italy